CLINICAL TRIAL: NCT05586399
Title: The Effect of Maximal Strength Training on Lung Function in Patients With COPD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Molde University College (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NA -COPD
Record Dates: First submitted 2022-09-06; First posted 2022-10-19 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-09

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Strength training; Lung function; Quality of life
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Pre-test 4 weeks before the intervention period (Subjects functioning as their own control), tests at baseline and 4 weeks after the intervention period.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise intervention (Experimental): Participants performing a rehabilitation program for 5 times a week in a total of 4 weeks in one of two rehabilitation centers in Trondheim, Norway. The aim is to perform a total of 20 maximal strength training interventions supervised by one or more health professionals. Maximal strength training will be performed with 4 repetitions and 4 series at 90-95% of one repetition maximum.
  Interventions: Behavioral: Maximal strength training in COPD

INTERVENTIONS:
Behavioral: Maximal strength training in COPD — Participate in a rehabilitation program for 4 weeks, with exercise 5 times a week. Supervised maximal strength training in a leg press machine for a total of 20 exercise sessions. Patients will participate in rehabilitation in one of two rehabilitations centers in Trondheim, Norway.

SUMMARY:
The purpose of this study is to investigate the effect on maximal strength training on muscle function, lung function and quality of life for patients diagnosed with COPD grade II-III (Gold scale). Each patient will complete a total of 20 exercise session participating in a rehabilitation program for 4 weeks. Physiological and functional testing will be performed 4 weeks before the training intervention, at baseline and after the intervention period.

DETAILED DESCRIPTION:
COPD is a group of diseases which affect the pulmonary system and leads to airflow restrictions and breathing difficulty. Other healthcare related problems, such as chronic inflammation, reduced muscle function, anxiety, depression and cardiovascular diseases are often seen in patients who are diagnosed with COPD.

Frequent participation in physical activity has been shown to improve the general public health, and serve as a prevention for development of various chronic diseases. Physical activity has at the same time been shown to be effective in treatment of both pulmonary and cardiovascular diseases. It also has the potential to reduce the need for health services, and can replace or reduce the need for medicinal treatments.

In this study we are want to investigate the effect of maximal strength training in COPD patients grade II-III on both muscle function and lung function. Maximal strength training (MST) have previously been shown as a superior intervention to achieve increased 1RM and fast development of power, also known as rate of force development (RFD). Lung function in COPD patients has been shown in previous research to be improved following maximal strength training.

The participants will partake in a total of 20 MST interventions during a rehabilitation period of 4 weeks. The sessions will be distributed five times a week located in two different Rehabilitation Centers in Trondheim, Norway. The strength training will be performed in groups, supervised by one or more coworkers in the project. MST will be performed with 4 series of 4 RM in a horizontal leg press machine, supervised by a coworker in the project. As part of the rehabilitation program, participants will also perform endurance training parallell to the MST sessions.

The participants will function as their own control group in the project. They will participate in a pre-test 4 weeks before the intervention period. After the pre-test they will be instructed to live as usual for the next 4 weeks. They will then start the intervention period, with tests performed at start and end of the period.

Both subjective and objective measurements will be performed 4 weeks before, at baseline and after the intervention period. All physiological tests will be completed during the same day. A standardized work economy test on a treadmill will be used in assessment of endurance capacity, with an expected duration of 4 minutes. The work economy test will be followed by a standardized graded test of maximal oxygen consumption, with a maximal duration of 10 minutes. Both endurance tests will be performed on a treadmill, with continuous heart rate monitoring. Approximately 5-10 minutes after finishing the endurance tests, a test of maximal dynamic strength will be performed (1RM test). The test will be performed in a horizontal leg press machine. After three submaximal warm-up sets, the load will be gradually increased until the participant fails to perform the test. Duration of rest periods between sets will be standardized to 3 minutes. Rate of force development will also be assessed, with the use of a force plate in the same horizontal leg press machine. There will also be performed functional tests (6 minute walk test, Timed Up and Go and stair climb test). All participants will also answer standardized questionnaires regarding health related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* COPD-diagnosis grade II-III (Gold Classification)
* Patients in one of two rehabilitation centres in Trondheim, Norway.
* Must be able to perform the test procedures walking or running on a treadmill.
* Must participate in at least 18 of the 20 planned training sessions.

Exclusion Criteria:

* Other pulmonary disease than COPD
* Diabetes mellitus or other metabolic diseases
* Use of corticosteroids the last 6 weeks
* Pulmonary infection the last 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-11-15 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Maximal Strenght | 4 weeks before the intervention, at baseline and after 20 training sessions during 4 weeks weeks of rehabilitation.
  Measured in 1 repetition maximum (kg) in leg press.
Change in Rate of Force Development | 4 weeks before the intervention, at baseline and after 20 training sessions during 4 weeks weeks of rehabilitation.
  Measured in Newton using a force plate
Change in Forced Expiratory Volume (FEV1) | 4 weeks before the intervention, at baseline and after 20 training sessions during 4 weeks weeks of rehabilitation.
  Measured using spirometry as the maximal volume of air (liter) exhaled in the first second of expiration
Change in Peak Expiratory Flow (PEF) | 4 weeks before the intervention, at baseline and after 20 training sessions during 4 weeks weeks of rehabilitation.
  Measured using spirometry as the maximal speed of expiration (Measured as liter/min)
Change in Work Economy | 4 weeks before the intervention, at baseline and after 20 training sessions during 4 weeks weeks of rehabilitation.
  Measured using CPET walking on a treadmill at a standardized speed and incline (Measured as VO2 ml/kg/min)
Change in Maximal Oxygen Consumption | 4 weeks before the intervention, at baseline and after 20 training sessions during 4 weeks weeks of rehabilitation.
  Measured using CPET in maximal test walking until exhaustion(Measured as VO2 ml/kg/min)
Change in Stair Climbing-test | 4 weeks before the intervention, at baseline and after 20 training sessions during 4 weeks weeks of rehabilitation.
  Measured in seconds as the average of two attempts
Change in Timed up and Go-test | 4 weeks before the intervention, at baseline and after 20 training sessions during 4 weeks weeks of rehabilitation.
  Measured in seconds as the average of two attempts
Change in 6 Minutes Walk Test | 4 weeks before the intervention, at baseline and after 20 training sessions during 4 weeks weeks of rehabilitation.
  Measured in meters

SECONDARY OUTCOMES:
Changes in health-related quality of life - Norwegian RAND36 | 4 weeks before the intervention, at baseline and after 20 training sessions during 4 weeks weeks of rehabilitation.
  Questionnaire scoring on a 0-100 scale with higher scores identifying better outcomes
Changes in health-related quality of life - Hospital and Anxiety Score (HADS) | 4 weeks before the intervention, at baseline and after 20 training sessions during 4 weeks weeks of rehabilitation.
  Questionnaires - Change in total score from 0-21 where higher score may indicate anxiety and/or depression
Changes in health-related quality of life - International physical activity questionnaire (IPAQ) | 4 weeks before the intervention, at baseline and after 20 training sessions during 4 weeks weeks of rehabilitation.
  Questionnaires - Change in MET-minutes of physical acitivity a week with higher score identifying better outcomes
Changes in health-related quality of life - EQ-5D-5L | 4 weeks before the intervention, at baseline and after 20 training sessions during 4 weeks weeks of rehabilitation.
  Questionnaires - Change in health state from level 1-5 with lower level identifying better outcomes
Changes in health-related quality of life - Visual Analogue Scale (VAS) | 4 weeks before the intervention, at baseline and after 20 training sessions during 4 weeks weeks of rehabilitation.
  Questionnaires - Units on a Scale from 0-10 cm with lower score identifying better outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Jan Helgerud, PhD, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- My Workout - Medical Rehabilitation Clinic, Trondheim, Norway